CLINICAL TRIAL: NCT05579093
Title: Clinical Investigation of an Eye-Tracking Device as a Predictor of Delirium in the Recovery Room After Surgery With General Anesthesia
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAT9610; IRB00103151 (Other: Emory)
Record Dates: First submitted 2022-05-23; First posted 2022-10-13 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Delirium
Keywords: Neurotrack™
MeSH Terms: conditions — Delirium | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Cognitive test + Pupillary measure — Patients will be put into a quiet room with a computer and a webcam for a five minute assessment with the NeuroTrack™ testing. Study personnel will stay in the room, and be available for answering questions about using the online testing tool.
  After Neurotrack, pupillary responses will be recorded with the pupillometer with the PLR -3000TM. In brief, an eye cup attached to a pupillometer will be placed over one eye to allow measurement of the pupillary response to light. Once the eye cup is properly positioned, the reading takes approximately 5 seconds, after which time the eye cup will be removed. The reading will then be taken in the contralateral eye.

SUMMARY:
Neurotrack™ is an FDA-approved device for measuring and tracking cognitive decline, as may occur with age-related cognitive decline and Alzheimer's disease. The device uses a webcam (World Wide Web enabled camera) to assess eye-tracking as the subject views black-and-white images on the computer screen. The test takes less than 5 minutes to complete. This study will examine the feasibility and utility of pre-operative assessment of cognition using Neurotrack™ technology. The predictive value of Neurotrack™ will be compared to our previous work using pupillometry. The primary outcome is a measure of delirium in the recovery room and secondary outcomes include total length of stay, intensive care unit (ICU) length of stay, and readmissions within 30 days of surgery.

DETAILED DESCRIPTION:
How the brain restores baseline consciousness at the end of a perioperative anesthetic is not known. However, it is becoming increasingly evident that arousal after sleep, coma, or anesthesia is an active process, not a passive process relying on simple clearance of anesthetic drugs. Insight into the specific sequence of brain circuit activation and inactivation during the end of an anesthetic may not only lead to an understanding of anesthetic emergence but provide important information for the potential long-term consequences of anesthetic drugs (anesthetic neurotoxicity, and the role of anesthetic drugs in delirium and dementia). The possibility of anesthesia causing harm to the brains of our patients is a controversy that has received a lot of attention from anesthesiologists, surgeons, and patients alike. The investigators' approach is to determine if techniques based on eye movements and/or pupillometry can predict and guide the post anesthesia management of delirium.

The conventional pupillary exam involves assessment of pupil size, shape, symmetry, and reactivity to light. Mechanistically, the pupillary light reflex involves the retina, cranial nerve II and III, pretectal nucleus in the midbrain, Edinger-Westphal nuclei, and the ciliary ganglion. With the use of an automated pupillometer, the pupillary response to light can also be quantified with measures of maximal diameter, latency, constriction velocity, minimal diameter, and dilation velocity. Beyond the reliability and accuracy that the device affords, pupillometry may have other utilities, potentially predicting postoperative delirium, episodes of intracranial hypertension, and even supratentorial herniation.

On the other hand, smooth pursuit involves conjugate eye movements that are required to maintain an object in motion on the fovea. The mechanism is quite complex, involving the lateral geniculate nucleus, primary visual cortex, middle temporal visual cortex, frontal pursuit area, superior colliculus, several pontine nuclei, the cerebellum, and nuclei of cranial nerves III, IV, and VI. It should not be surprising that cortical atrophy that occurs with normal aging or a dementing process may alter eye movements. The utility and relationship of pupillometry and Neurotrack™, alone and in combination with intraoperative electroencephalogram (EEG), is of immense interest. Prediction of post-operative delirium and cognitive decline with simple non-invasive means would be a significant clinical advancement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater
2. Any American Society of Anesthesiologists (ASA) classification
3. Scheduled elective surgery with general anesthesia. Extubation, and emergence anticipated in the operating room and recovery in the post-operative care unit (PACU).

Exclusion Criteria:

1. Cardiac surgery (on or off cardiopulmonary bypass).
2. Intracranial neurosurgery
3. Surgery involving the eye, eyebrow, forehead, or frontal scalp near the eyes
4. Emergency surgery
5. Monitored Anesthesia Care (i.e., regional anesthesia alone without anticipated plans for general anesthesia)
6. Poor health literacy ("How confident are you filling out medical forms by yourself?")
7. Endotracheal intubation maintained upon leaving operating room
8. Direct admission to ICU due to foreseen or unforeseen circumstances

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sign-up for the protocol will be based upon a review of the preoperative and pre-op clinic schedules, a recommendation from operating room physicians or referral from preoperative anesthesia consultant at the conclusion of their preoperative clinic visit. A clinical research coordinator or other research personnel is available to answer questions and obtain informed consent from the patient. It will be made clear to the patient that study participation is optional and that they can "opt out" at any time even if they have signed a consent form.
  We intend on enrolling male and female patients that meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of delirium | Up to 2 years
  Prevalence of delirium in in the post anesthesia care unit (PACU) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Garcia, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided